CLINICAL TRIAL: NCT01721668
Title: Examination of Therapeutic Intervention Methods on the Brain Recovery
Brief Title: Improving Arm and Hand Functions in Chronic Stroke (CIHR 2012-2015)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Deirdre Dawson, Dr. Deirdre Dawson, Senior Scientist Rotman Research Institute, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB1213
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSR - Music Supported Rehabilitation (Experimental): Behavioral: Music Supported Rehabilitation
  Interventions: Behavioral: Music Supported Rehabilitation
- CU/ET (Active Comparator): Experimental: CU/ET (Conventional Upper Extremity Therapy)
  Interventions: Behavioral: Conventional Upper Extremity Therapy

INTERVENTIONS:
Behavioral: Music Supported Rehabilitation — Music Supported Rehabilitation -using musical exercises to improve hand and arm motor functioning.
  Arms: MSR - Music Supported Rehabilitation
Behavioral: Conventional Upper Extremity Therapy — -GRASP (Graded Repetitive Arm Supplementary Program-developed Janice Eng, PhD, PT/OT Jocelyn Harris, PhD, OT, Andrew Dawson, MD, FRCP, Bill Miller, PhD, OT) protocol will be used to improve arm and hand function in people living with stroke.
  Arms: CU/ET

SUMMARY:
Improving arm and hand function after stroke has been difficult to achieve within the rehabilitation service provided in the acute stage often due to the limited resource in health care. While spontaneous recovery plateaus after 6 months, the prolonged disability affects quality of life and social participation in stroke survivors. This study is aimed at improving chronic motor impairment arm and hand impairment by providing the intervention with intensive training schedule. This study will compare two types of rehabilitation intervention using a randomized controlled trial. Measurements also will be taken on various brain functions non-invasively to help discover how each of the intervention strategies works differently to repair the brain.

DETAILED DESCRIPTION:
After unilateral stroke, incomplete recovery of arm and hand movement is common and its long-lasting negative effects include increased care giving costs and overall reduced quality of life. Recent evidence suggests that a novel behavioral intervention could improve motor functions in sub-acute patients with added benefits in cognitive and brain functions. However few studies have addressed whether chronic stage patients can also benefit from the intervention and how brain plasticity works over the course of rehabilitation. This study will investigate the benefits of two types of intervention methods that are extendable for community-based intervention services in the future. It also will examine changes in integrity of motions before and after the intervention. Further comparisons between brain functions and structure will be made using magnetoencephalography (MEG) and magnetic resonance imaging (MRI), non-invasively. These behavioural and physiological measures will inform the mechanisms of stroke recovery and training.

ELIGIBILITY:
Inclusion Criteria:

* post-acute stroke patients with unilateral first-time MCA stroke sustained . (more than 6 months ago prior to the enrolment to the study).
* Patients' residual motor impairments in the affected hand and arm should be greater than stage 3 on the Chedoke McMaster scale.

Exclusion Criteria:

* Patients with moderate apraxia, aphasia or dementia, and patients with severe sensory loss in the paretic hand, severe language-communication disability, posture problems, involuntary movements, high-blood pressure, depression or other psychological disorders, metal in body that interferes with MEG and MRI measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in performance on Action Research Arm Test | Baseline, post-5-weeks, post-10-weeks, and 4-month-follow-up
  Changes in performance from baseline to post-intervention at 5 weeks, to post-intervention at 10 weeks, and to follow-up at 4 mos will be measured.
Change in performance on Chedoke Arm and Hand Inventory | Baseline, post-5-weeks, post-10-weeks, and 4-month-follow-up
  Changes in performance from baseline to post-intervention at 5 weeks, to post-intervention at 10 weeks, and to follow-up at 4 mos will be measured.
Change in status on Stroke Impact Scale | Baseline, post-5-weeks, post-10-weeks, and 4-month-follow-up
  Changes in performance from baseline to post-intervention at 5 weeks, to post-intervention at 10 weeks, and to follow-up at 4 mos will be measured.

SECONDARY OUTCOMES:
Brain structure | Pre, post-5-weeks, post-10-weeks, and 4-month-follow-up
  Structural MRI
Brain Function | Baseline, post-5-weeks, post-10-weeks, and 4-month-follow-up
  Brain functions related to sensory and motor systems assessed by MEG

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre R Dawson, PhD, Principal Investigator — Baycrest; Bernhard Ross, PhD, Principal Investigator — Baycrest; Takako Fujioka, PhD, Principal Investigator — Stanford University
Locations (1):
- Baycrest Centre for Geriatric Care, Toronto, Ontario, Canada